CLINICAL TRIAL: NCT03854461
Title: The Efficacy of Individualized Dietary Advice in Improving Diet Quality and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: University College Dublin (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK120870-01
Record Dates: First submitted 2019-02-19; First posted 2019-02-26 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
Keywords: individualised dietary advice; biomarkers; diet quality; cardiometabolic health
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomised parallel group dietary intervention: two group.
Who Masked: Outcomes Assessor
Masking Description: All outcomes will be conducted blind, including the primary outcome (diet quality score), laboratory analysis and cardiometabolic health marker assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational material (Active Comparator): Participants will be given written educational material to encourage dietary change towards a better quality diet. Educational material will be adapted from resources used in previous dietary intervention studies.
  Interventions: Behavioral: Educational material
- Personalised dietary advice and educational material (Experimental): Participants will also be given the educational material, but will be encouraged to make dietary change using individualized recommendations incorporating food markers of specific components of a high quality diet. Food markers of diet quality will be used to develop an algorithm to deliver personalized dietary advice. Based on biomarker data, a system of categorization of biomarker status will be developed, alongside dietary advice related to this biomarker categorization, and decision trees created, as previously described in the Food4Me study, to ensure standardized delivery of advice within this intervention arm.
  Interventions: Behavioral: Personalised dietary advice and educational material

INTERVENTIONS:
Behavioral: Personalised dietary advice and educational material — As within arm/group description
  Arms: Personalised dietary advice and educational material
Behavioral: Educational material — As within arm/group description
  Arms: Educational material

SUMMARY:
This study is a a randomized controlled parallel group dietary intervention conducted over six months in participants at high risk of cardiovascular disease living in Ireland (North and South) to evaluate the efficacy of individualized dietary advice incorporating biomarker profiles in improving diet quality and cardiometabolic outcomes.

DETAILED DESCRIPTION:
Study design: a randomized controlled parallel group dietary intervention will be conducted over six months in participants at high risk of CVD living in Ireland (North and South) to evaluate the efficacy of individualized dietary advice incorporating biomarker profiles in improving diet quality and cardiometabolic outcomes.

Population and recruitment

Population characteristics: Participants will be at high risk (>20% over 10 years) of developing CVD. Established recruitment mechanisms, used in several previous and ongoing dietary intervention studies, from general practices, hospital outpatient clinics, and from the general population (via press release, radio interviews, poster placement) will be utilized.Recruitment will take place over an 18 month period.

Inclusion criteria: Participants will be considered eligible to enroll in the study if they are overweight (BMI >27 and ≤ 45 kg/m2), have low Prime Diet Quality Score (PDQS <15)27 and a combination of risk factors which places them at high total risk (estimated multifactorial CVD risk ≥ 20% over ten years) of developing atherosclerotic CVD for the first time.

Exclusion criteria: Participants will be ineligible to enroll in the study if they have established diabetes mellitus, CVD or a medical condition or dietary restriction(s) that would substantially limit their ability to complete the study requirements, have an excessive alcohol consumption (>28 Units/week for men or >21 Units/week for women), have a low predicted likelihood to change dietary habits or are unable to provide informed consent.

Randomization: A personal health and medical history questionnaire, together with Joint British Societies CVD risk prediction charts and an assessment of participant's baseline PDQS using a 42-item questionnaire will be used to assess eligibility. This questionnaire is validated in the US, but will be validated in the Irish population. Those eligible and willing to take part will give informed written consent, and will be randomized (randomization scheme generated using www.randomization.com with random block sizes and research staff administering the randomization or conducting endpoint assessment blinded) to either an education only intervention or individually tailored food marker-based dietary advice.

The intervention will take place over a six month period. Participants will be interviewed towards the end of the intervention (for those in individually tailored support arm), or at drop-out (for all participants who drop out), to elicit their views on the intervention.

Dietary intervention: Participants will be randomized to one of two groups:

1. Control - participants will be given written educational material to encourage dietary change towards a better quality diet. Educational material will be adapted from resources used in previous dietary intervention studies.
2. Personalized dietary advice - participants will also be given the educational material, but will be encouraged to make dietary change using individualized recommendations incorporating food markers of specific components of a high quality diet. Food markers of diet quality will be used to develop an algorithm to deliver personalized dietary advice. Based on biomarker data, a system of categorization of biomarker status will be developed, alongside dietary advice related to this biomarker categorization, and decision trees created, as previously described in the Food4Me study, to ensure standardized delivery of advice within this intervention arm.

The dietary advice will be delivered via email and online, with monthly contact and the messages being reinforced during each direct contact with the study team for outcome assessment. Therefore frequency and duration of contact will be similar in both intervention groups.

Outcome measures: Outcomes will be assessed during a clinic visit at 0, 3 and 6 months, and will include dietary intake, anthropometry, other lifestyle behaviors, blood pressure, biological sample collection for nutritional status biomarker and health biomarker analysis, as well as fecal samples for metagenomic and transcriptomic profiling. Outcome data will be collected using the following methodology:

* Demographic/lifestyle information (e.g., alcohol consumption, medication use).
* Dietary intake using an online version of the PDQS. This will also be assessed six months after the intervention completes, to determine whether the intervention influences longer term adherence to a better quality diet.
* Physical activity using an objective physical activity monitor.
* Anthropometric data (weight and height measured using calibrated scales and stadiometer respectively, waist and hip circumference); body composition by bioelectrical impedence (Bodystat 1500).
* Blood pressure will be measured twice from the right arm, using an automated Omron sphygmomanometer, with the participant sitting quietly for at least five minutes.
* Fasting blood samples will be drawn from the antecubital vein and immediately separated into plasma/serum for the proposed assays detailed below. It will be stored at -70°C until analysis.
* Fasting morning urine sample stored at -70ºC until analysis.
* In a subset of participants (n=70, 35 in each arm), stool samples will be collected at baseline and the end of intervention for the analysis of changes in gut microbiota composition and functionality, as previously described.

Laboratory methodology: All methods are in routine use in participating laboratories and are performed with careful attention to quality control and with participation in external quality control schemes where available. All laboratory analysis will be conducted blind, i.e. the analyst will not know to which intervention the participant has been assigned.

Biomarkers of cardiometabolic risk: Serum lipids (total cholesterol, HDL-C, and TG) and whole blood HbA1c will be assessed by enzymatic assays (Randox Ltd, Crumlin, NI and Glen Bio, Antrim, NI) on an I-Lab 600 auto-analyzer. LDL-C will be calculated.

Biomarkers of diet quality: the following biomarkers will be used to assess nutritional status response to the dietary intervention: red meat - methylhistidines and carnosine; white meat - TMAO, guanidoacetate, anserine; fruit and vegetables -- proline betaine, isothiocyanates, S-methyl-L-cysteine sulfoxide, and tartaric acid; wholegrains - alkylresorcinols; coffee - phenolic acids, N-methylpyridinium, trigonelline, 2-furoylglycine; SSBs -- formate, citrulline, taurine, and isocitrate)red meat- methylhistidines; oily fish- omega-3 index; fruit and vegetables- total carotenoids and proline betaine; wholegrain- alkylresorcinols.

Gut microbiota composition and functionality: Sample handling and nucleic acid purifications will be performed following an established protocol.166 Illumina DNA-seq libraries with fragment length of ~300 bp will be generated, with Pippen prep size selection. For RNA-seq, 5ug of RNA will be enriched for mRNA and subjected to strand-specific cDNA synthesis using established protocols. Paired-end sequencing (e.g. 150x150 nt) will be performed on the Illumina HiSeq platform.

Primary Outcome: Change in Prime Diet Quality Score.

Secondary Outcomes:

1. Change in markers of cardiometabolic risk, including blood pressure, lipid profile, HbA1c, body weight.
2. Change in biomarkers of diet quality
3. Gut microbiota composition and functionality (to be conducted in a subset).

Power calculation: Sample size calculations will be confirmed during the validation of the PDQS within an Irish population. However, based on published US data, with a standard deviation (SD) of PDQS of 2.3, and an assumption of a difference in increase in PDQS of 5 between the personalized dietary advice and control groups then, if there are 60 participants in each group, the study would have over 90% power to detect this difference in mean PDQS as statistically significant, at the α=0.05 level. A total of 134 participants will be recruited to allow for approximately 10% drop-out. For the health outcomes, and, based on what was observed in a dietary intervention based on improving diet quality in similar high CVD risk participants, if there are 60 participants in each group, and it is assumed that (i) the SD of the change in diastolic blood pressure (DBP) is 9 mmHg at the end of the study; (ii) a difference in DBP of 4.5 mmHg between the individualized dietary advice and control groups; then the study would have 80% power to detect, as statistically significant at the 5% level, these differences in mean change between the two groups. The investigators will have similar levels of power (~80%) to detect effect sizes of similar magnitude in total cholesterol, HbA1c and body weight. The analysis of gut microbiota composition and functionality will be exploratory in nature.

Data analytical strategy: The repeated end-point measures generated by the study design will be analyzed with techniques appropriate for longitudinal data using the xt panel study procedures available in Stata release 11 (College Station, TX). Initial examination of the correlation structure of the repeated measures will help guide model fitting. The influence of the dietary intervention under study will be assessed by comparing the means of changes in measurements from baseline to 6 months between the biomarker-based individually tailored advice and education only groups. This difference in means will provide an estimate of the effect of intervention and 95% confidence limits will be calculated to indicate its precision. If appropriate, measurements will be logarithmically transformed prior to analysis and interpretation will be made in ratio terms on the original scale.

ELIGIBILITY:
Participants will be at high risk (>20% over 10 years) of developing CVD.

Inclusion Criteria:

Participants will be considered eligible to enroll in the study if they are:

1. overweight (BMI >27 and ≤ 45 kg/m2),
2. have low Prime Diet Quality Score (PDQS <15) and
3. have a combination of risk factors which places them at high total risk (estimated multifactorial CVD risk ≥ 20% over ten years) of developing atherosclerotic CVD for the first time.

Exclusion Criteria:

Participants will be ineligible to enroll in the study if they have:

1. established diabetes mellitus, CVD or a medical condition or dietary restriction(s) that would substantially limit their ability to complete the study requirements,
2. have an excessive alcohol consumption (>28 Units/week for men or >21 Units/week for women),
3. have a low predicted likelihood to change dietary habits
4. are unable to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Public Health, Institute of Clinical Sciences A, Queen's University Belfast, Grosvenor Road, Royal site. Road, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
At early planning stage of study - undecided.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between December 2021 and November 2022 at both Queen's University Belfast, Northern Ireland and University College Dublin, Republic of Ireland sites.
Pre-assignment Details: As n=12 participants who were enrolled onto the study were not contactable afterwards to arrange baseline (Month 0) study visits, n=162 participants in total were enrolled to account for losses identified early in data collection process before baseline visit. N=150 completed baseline (Month 0) visits but n=1 participant was discovered to be ineligible at baseline visit and was removed. Therefore n=149 completed baseline visits and were randomised.
Period: Overall Study
Arm/Group | Educational Material | Personalised Dietary Advice and Educational Material
Started | 74 | 75
Completed | 63 | 56
Not Completed | 11 | 19

BASELINE CHARACTERISTICS:
Population: N=1 participant was deemed ineligible at baseline study visit and was removed-they had withheld relevant information at screening.
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Material | Personalised Dietary Advice and Educational Material | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (continuous), in years
  years | 48.4 (12.9) | 50.3 (11.2) | 49.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 55 | 106
  Male | 23 | 20 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Prime Diet Quality Score [Mean (Standard Deviation); unit: PDQS score] — Diet Quality Assessment determined via mean Prime Diet Quality Score (range 0-42)
  PDQS score | 14.9 (3.9) | 16.1 (4.6) | 15.5 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean Change in Prime Diet Quality Score Between Groups Between Months 0 and 6
Description: Dietary quality will be assessed using an online version of the Prime Diet Quality Score (PDQS). Foods are classified as healthy and unhealthy. Points are assigned according to the following criteria: 0-1 serving/wk (0 point) compared with 2-3 servings/wk (1 point) compared with ≥4 servings/wk (2 points) for the healthy food groups. Scoring is reversed and points deducted for the unhealthy food groups. Points for each food group are summed to give an overall score. The PDQS has 21 food groups and ranges from 0 to 42 total score (scores on a scale), with a higher score indicating a better diet quality.
Time Frame: Baseline and six months
Population: Primary outcome was assessed via questionnaire. At Month 6 some participants completed questionnaire only (including primary outcome) but not visits (secondary outcomes; whilst some participants completed visits only (secondary outcomes) but not questionnaires (primary outcome).
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Difference in Mean Change Between Groups (Xtreg) (95% CI): Dietary intake was assessed using an online version of the Prime Diet Quality Score (PDQS). Foods were classified as healthy and unhealthy. Points were assigned according to the following criteria: 0-1 serving/wk (0 point) compared with 2-3 servings/wk (1 point) compared with ≥4 servings/wk (2 points) for the healthy food groups. Scoring will be reversed and points deducted for the unhealthy food groups. Points for each food group will be then summed to give an overall score. The PDQS has 21 food groups and ranges from 0 to 42 total points.
  Difference in mean change in PDQS between education and comparator groups between Months 0 and 6 was the primary outcome.
Arm/Group | Difference in Mean Change Between Groups (Xtreg) (95% CI)
Number analyzed (Participants) | 119
Units on a scale | 1.22 [-0.51 to 2.95]

2. Secondary Outcome: Alcohol Consumption
Description: Questionnaire to assess number of units consumed weekly
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

3. Secondary Outcome: Medication Use
Description: Questionnaire to assess usual medication use (drug name, dose and frequency of use)
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

4. Secondary Outcome: Physical Activity
Description: Physical activity using an accelerometer; data to be used will be total step count
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

5. Secondary Outcome: Anthropometric Data - Weight
Description: Weight will be measured in kg using calibrated scales.
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

6. Secondary Outcome: Anthropometric Data - Waist to Hip Ratio
Description: Waist and hip circumference will be measured in cm according to standardised operating procedures using a tape measure.
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

7. Secondary Outcome: Anthropometric Data - Height
Description: Height will be measured in metres using a stadiometer.
Time Frame: Baseline and six months
Reporting Status: Not Posted

8. Secondary Outcome: Anthropometric Data - Body Composition.
Description: Body composition (% body fat) will be measured using bioelectrical impedence (Bodystat 1500).
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

9. Secondary Outcome: Blood Pressure
Description: Blood pressure will be measured twice from the right arm, using an automated Omron sphygmomanometer, with the participant sitting quietly for at least five minutes.
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

10. Secondary Outcome: Biomarkers of Cardiometabolic Risk
Description: Serum lipids (total cholesterol, HDL-C, and TG) and whole blood HbA1c will be assessed by enzymatic assays (Randox Ltd, Crumlin, NI and Glen Bio, Antrim, NI) on an I-Lab 600 auto-analyzer. LDL-C will be calculated.
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

11. Secondary Outcome: Biomarkers of Diet Quality
Description: The following biomarkers will be used to assess nutritional status response to the dietary intervention: red meat - methylhistidines and carnosine; white meat - TMAO, guanidoacetate, anserine; fruit and vegetables -- proline betaine, isothiocyanates, S-methyl-L-cysteine sulfoxide, and tartaric acid; wholegrains - alkylresorcinols; coffee - phenolic acids, N-methylpyridinium, trigonelline, 2-furoylglycine; SSBs -- formate, citrulline, taurine, and isocitrate) red meat- methylhistidines; oily fish- omega-3 index; fruit and vegetables- total carotenoids and proline betaine; wholegrain- alkylresorcinols.
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

12. Secondary Outcome: Gut Microbiota Composition (Subset of Participants Only)
Description: Sample handling and nucleic acid purifications will be performed following an established protocol. Illumina DNA-seq libraries with fragment length of ~300 bp will be generated as previously described, with Pippen prep size selection. For RNA-seq, 5ug of RNA will be enriched for mRNA and subjected to strand-specific cDNA synthesis using established protocols. Paired-end sequencing (e.g. 150x150 nt) will be performed on the Illumina HiSeq platform.
Time Frame: Baseline and six months
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 1 year.
Arm/Group | Personalised Dietary Advice and Educational Material | Educational Material
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 0/75 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03854461/Prot_SAP_000.pdf